CLINICAL TRIAL: NCT01532310
Title: WEUKBRE6076: Belimumab (BENLYSTA) Pregnancy Registry Protocol
Brief Title: Belimumab (BENLYSTA®) Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: 114256; WEUKBRE6076 (Other: GSK)
Record Dates: First submitted 2012-02-02; First posted 2012-02-14 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; belimumab; pregnancy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant women taking belimumab: Any women with belimumab exposure within the 4 months prior to and/or during pregnancy
  Interventions: Drug: belimumab
- Infants: Infants through the first year of life whose mothers were exposed to belimumab during pregnancy
  Interventions: Drug: belimumab

INTERVENTIONS:
Drug: belimumab — Belimumab is a recombinant, human, IgG1λ monoclonal antibody for the treatment of systemic lupus erythematosus

SUMMARY:
This global Belimumab Pregnancy Registry will collect prospective data on pregnancies and pregnancy outcomes on a voluntary basis in women with systemic lupus erythematosus (SLE) who have received commercially supplied belimumab within the 4 months prior to and/or during pregnancy. The registry will also evaluate outcomes of infants born to mothers who were exposed to belimumab within the 4 months prior to and/or during pregnancy. This registry will add to the current clinical experience with belimumab and will complement reproductive data from animal toxicology studies. It will also assist clinicians in weighing the potential risks against the benefits of treatment for individual patients with SLE. GlaxoSmithKline (GSK) will sponsor the Belimumab Pregnancy Registry in countries where it holds Marketing Authorization.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women containing sufficient evidence to confirm that exposure to commercially supplied belimumab occurred within the 4 months prior to and/or during pregnancy
* Pregnant women with sufficient information to classify the pregnancy as prospective or retrospective (ie,whether the outcome of pregnancy was known at the time of first contact with the registry)
* Pregnant women with full contact information to allow for follow-up (name, address, telephone number/email address) and contact information for applicable HCPs if initial reporter is the pregnant woman
* Consent provided by the pregnant woman for her participation and assent for participation of her infant.

Exclusion Criteria:

* Reported cases that do not meet the minimum inclusion criteria for registry enrollment will be ineligible for inclusion in the registry

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with SLE who have been exposed to commercially supplied belimumab within the 4 months prior to and/or during pregnancy will be eligible to participate in the registry as well as their infants.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Birth defects | Up to one year after birth
  The registry will define and code birth defects with criteria specified by Centers for Disease Control and Prevention (CDC)'s Metropolitan Atlanta Congenital Defects Program (MACDP)

SECONDARY OUTCOMES:
Other pregnancy outcomes | At birth
  Other pregnancy outcomes including spontaneous miscarriage, live birth (including pre-term birth and small for gestational age), stillbirth, and elective termination
Infant outcomes | Up to 1 year after birth
  Serious and/or clinically significant infections

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- GSK Investigational Site, Wilmington, North Carolina, United States
- GSK Investigational Site, Innsbruck, Austria
- GSK Investigational Site, Liège, Belgium
- GSK Investigational Site, Québec, Quebec, Canada
- GSK Investigational Site, Paris, France
- GSK Investigational Site, Düsseldorf, Germany
- GSK Investigational Site, Tel Litwinsky, Israel
- GSK Investigational Site, Pisa, Italy
- GSK Investigational Site, Almada, Portugal
- GSK Investigational Site, Bilbao, Spain
- GSK Investigational Site, Stockholm, Sweden
- Switzerland (3):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich

REFERENCES:
- [Background] Juliao P, Wurst K, Pimenta JM, Gemzoe K, Landy H, Moody MA, Tilson H, Covington D, Moore T, Marino R, Gilbride J, Liu A, Meizlik P, Petri M. Belimumab use during pregnancy: Interim results of the belimumab pregnancy registry. Birth Defects Res. 2023 Jan 15;115(2):188-204. doi: 10.1002/bdr2.2091. Epub 2022 Sep 30. PMID 36177676
- See also: Belimumab pregnancy registry/GlaxoSmithKline pregnancy registries — http://pregnancyregistry.gsk.com/belimumab.html